CLINICAL TRIAL: NCT07298564
Title: Assessment of the Effect of Magnesium and Levocarnitine Co-supplementation on Lipid Profile, Glycemic Control Indicators and Hirsutism in Women With Polycystic Ovarian Syndrome
Brief Title: Effect of Magnesium and Levocarnitine on Metabolic and Clinical Outcomes in Women With Polycystic Ovarian Syndrome (PCOS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Behnood Abbasi (Other)
Responsible Party: Sponsor-Investigator, Behnood Abbasi, Clinical Professor, Science & Research Islamic Azad University Branch Khozestan
Organization: Science & Research Islamic Azad University Branch Khozestan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.IAU.SRB.REC.1404.234
Record Dates: First submitted 2025-12-06; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome; Hyperandrogenism; Insulin Resistance; Dyslipidemia; Hirsutism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Insulin Resistance; Dyslipidemias; Hirsutism | interventions — Magnesium; Carnitine

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group interventional study designed to evaluate the effects of magnesium and levocarnitine co-supplementation on metabolic and clinical parameters in women with Polycystic Ovary Syndrome (PCOS). Participants will be randomly assigned to one of three parallel groups: (1) magnesium supplementation plus placebo levocarnitine , (2) levocarnitine and magnesium co-supplementation, or (3) placebo. The intervention period lasts 12 weeks, and outcomes include lipid profile, glycemic control, and hirsutism severity.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is designed as a triple-blind randomized controlled trial. Participants, care providers, and investigators responsible for data collection and intervention administration will be blinded to group allocation. Before the study, containers will be coded as A, B and C by a person other than the study researchers according the concealment rules .The supplements (magnesium, L-carnitine, and placebo) will be identical in appearance, taste, and packaging, and labeled with coded numbers by an independent pharmacist who is not involved in the study procedures or data analysis. Group codes will be kept sealed until the completion of data analysis. This approach ensures the concealment of allocation and minimizes performance and detection bias throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Magnesium 500 mg and Placebo Levocarnitine (Experimental): Magnesium 500Mg Oral Tablet and placebo matching Levocarnitine 1000 mg daily
  Interventions: Dietary Supplement: Magnesium 500 mg; Dietary Supplement: Placebo Levocarnitine
- Levocarnitine 1000 mg and Magnesium 500 mg (Experimental): Levocarnitine supplement 1000 mg daily, along with magnesium 500 mg daily in two divided doses of 250 mg
  Interventions: Dietary Supplement: Levocarnitine 1000 mg; Dietary Supplement: Magnesium 500 mg
- Placebo (Placebo Comparator): Placebo capsules matching magnesium and Levocarnitine for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium 500 mg — Participants will receive magnesium supplement 500 mg daily in two divided doses of 250 mg each for 12 weeks.
  Magnesium Placebo
  Arms: Magnesium 500 mg and Placebo Levocarnitine
Dietary Supplement: Levocarnitine 1000 mg — Participants will receive Levocarnitine supplement 1000 mg daily for 12 weeks.
  Arms: Levocarnitine 1000 mg and Magnesium 500 mg
Dietary Supplement: Placebo — Participants will receive placebo capsules matching magnesium and Levocarnitine for 12 weeks.
  Arms: Placebo
Dietary Supplement: Magnesium 500 mg — Participants will receive magnesium 500 mg daily in two divided doses of 250 mg each for 12 weeks.
  Arms: Levocarnitine 1000 mg and Magnesium 500 mg
Dietary Supplement: Placebo Levocarnitine — Participants will receive placebo matching Levocarnitine 1000 mg daily for 12 weeks.
  Arms: Magnesium 500 mg and Placebo Levocarnitine

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is one of the most common endocrine disorders among women of reproductive age and is associated with metabolic abnormalities such as insulin resistance, dyslipidemia, and hormonal imbalance, which may lead to infertility and hirsutism. Despite the availability of several pharmacological treatments, many therapies fail to effectively address the underlying metabolic and endocrine dysfunctions of PCOS. Magnesium and L-carnitine are two essential nutrients that may play a synergistic role in improving insulin sensitivity, glucose metabolism, and lipid profile, as well as reducing oxidative stress and androgen production in women with PCOS. This randomized, triple-blind, placebo-controlled clinical trial aims to evaluate the effects of co-supplementation with magnesium and L-carnitine on glycemic control indices, lipid profile, and hirsutism in women with PCOS. A total of 84 eligible women aged 19-65 years diagnosed with PCOS according to the Rotterdam criteria will be recruited from Shohada Tajrish Hospital, Tehran, Iran. Participants will be randomly assigned to one of three groups: (1) magnesium supplementation (500 mg/day, in two 250 mg doses) plus L-carnitine placebo, (2) L-carnitine supplementation (1000 mg/day) plus magnesium (500 mg/day), or (3) placebo control group. The intervention period will last 12 weeks. Physical activity information will be collected using short form of International Physical Activity Questionnaire (IPAQ) and demographic information through a general information questionnaire. In order to evaluate dietary intake of patients in terms of energy(kcal/(day), carbohydrate(gr/day), protein(gr/day), fat intake(gr/day), saturated fatty acids (SFA) (gr/day), monounsaturated fatty acids (MUFA) (gr/day), polyunsaturated fatty acids (PUFA)(gr/day), Vitamin E (mg/day), Vitamin C (mg/day), Beta-carotene (mg/day) and Vitamin A (mg/day), cupper intake (mg/day), selenium intake (mg/day), and zink intake (mg/day), 24-hr recalls will be completed by interviewing the patient for 3 days (two normal days and a weekend day). Weight will be measured with the minimum dress and without shoes by using a digital balance scale of 100 grams and height will be measured without shoes by meters mounted to the wall with an accuracy of 0.5 centimeters. Then the body mass index will be calculated by dividing the weight (kg) by the square of the height (m), waist circumference will be measured in the narrowest area between the lowest lumbar spine and the iliac bone (cm), systolic and diastolic blood pressure will be measured after 15 minutes of rest, twice using the mercuric barometric measure and the mean will be reported as individual blood pressure. The blood sample will be taken after 12 hours of overnight fasting in three groups for measuring Fasting Blood Sugar (FBS) (mg/dL), lipid profile (mg/dL), Hemoglobin A1c (HbA1C) (percentage), serum insulin concentration (µIU/ml) and insulin resistance. Insulin resistance will be calculated using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) formula, and hirsutism score (using the modified Ferriman-Gallwey method) will be assessed at baseline and post-intervention. At the end of the study, counting the remaining capsules, the patient's compliance rate will be evaluated, and patients who have consumed less than 90% of their capsules will be excluded from the analysis.

DETAILED DESCRIPTION:
This is a randomized, triple-blind, parallel clinical trial evaluates the effects of co-supplementation with Magnesium and Levocarnitine on metabolic and hormonal outcomes in women with Polycystic Ovary Syndrome (PCOS). Patients are randomly assigned into three groups and received magnesium supplementation (500 mg/day, in two 250 mg doses), L-carnitine supplementation (1000 mg/day), and placebo for 12 weeks. Then the body mass index, waist circumference, systolic and diastolic blood pressure, Fasting Blood Sugar (FBS), lipid profile, Hemoglobin A1c (HbA1C), serum insulin concentration and insulin resistance are measured; All assessments will be performed at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 65 years.
* Diagnosis of polycystic ovary syndrome (PCOS) according to the Rotterdam criteria.

Exclusion Criteria:

* Hypothyroidism
* Menopause
* Pregnancy or breastfeeding
* Renal (kidney) dysfunction
* Use of therapeutic vitamin or mineral supplements
* Liver diseases (e.g., grade 3 fatty liver, hepatitis, or cirrhosis)
* Psychiatric disorders such as bipolar disorder
* Neuromuscular diseases (e.g., myasthenia gravis, Parkinson's disease, multiple sclerosis, epilepsy, or muscular dystrophy)
* History of seizures
* Participants who become pregnant during the study or fail to comply with more than 20% of the study protocol will be withdrawn from the study

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of FBS | Baseline and 12 weeks after
  Fasting blood glucose concentration (mg/dl) (mg/dL)

SECONDARY OUTCOMES:
Change from Baseline of serum insulin | Baseline and 12 weeks after
  Serum insulin (µIU/mL)
Change from baseline of HbA1c | Baseline and 12 weeks after
Change from baseline of HOMA-IR | Baseline and 12 weeks after
  Calculated as [fasting glucose (mg/dL) × fasting insulin (µIU/mL) / 405]
Change from baseline of total cholesterol | Baseline and 12 weeks after
  Serum TC (total cholesterol) concentration (mg/dl)
Change from baseline of Triglyceride | Baseline and 12 weeks after
  Serum TG (triacylglycerol) concentration (mg/dl)
Change from baseline of low density lipoprotein cholesterol (LDL-Cholesterol) | Baseline and 12 weeks after
  Serum LDL concentration (mg/dl)
Change from baseline of high density lipoprotein cholesterol (HDL-Cholesterol) | Baseline and 12 weeks after
  Serum HDL concentration (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Tara Momeni, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: No